CLINICAL TRIAL: NCT03601741
Title: Use of Disposable Stethoscope Covers for Reduction of Stethoscope MRSA Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17-01633
Record Dates: First submitted 2018-05-02; First posted 2018-07-26 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: MRSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial Stethoscope Diaphragm Covers (Active Comparator)
  Interventions: Other: Daily Antimicrobial Stethoscope Diaphragm Cover; Other: Uncovered Stethoscopes
- Uncovered Stethoscopes (Active Comparator)
  Interventions: Other: Daily Antimicrobial Stethoscope Diaphragm Cover; Other: Uncovered Stethoscopes

INTERVENTIONS:
Other: Daily Antimicrobial Stethoscope Diaphragm Cover — Patients will receive package with instructions to use stethoscope cover, and are then instructed to switch in 7 days
Other: Uncovered Stethoscopes — Patients receive instruction to begin with no covers, and are then instructed to switch in 7 days

SUMMARY:
This is a prospective pilot study using a randomized, controlled, single blinded, crossover trial design, evaluating the effect of daily antimicrobial stethoscope diaphragm covers versus uncovered stethoscope. Stethoscopes will be cleaned Sani-cloth germicidal disposable wipes which are effective against MRSA. Each participant will then be randomly assigned to 7 days in either the intervention or the control arm. At the end of the 7 days participants stethoscopes will be cleaned again. This will be followed by another 7 days in the arm that they are not in during the first 7 days.

The primary endpoint is MRSA colony count from stethoscope diaphragms cultures at 7 days, focusing on the difference between the intervention and the control periods. The secondary endpoint is the rate of hospital acquired MRSA infection in patients treated by residents during each period.

ELIGIBILITY:
Inclusion Criteria:

* Internal Medicine Residents

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
MRSA colony count cultured from stethoscope diaphragms | 7 Days
  Total CFU of each selected pathogen at 7 days compared by paired Mann-Whitney U tests, with each patient serving as their own control

SECONDARY OUTCOMES:
Rate of hospital acquired MRSA infection in patients treated by participating residents | 14 Days
  Rates on nosocomial infection in each arm compared through use of Kaplan Meier curves

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Moussa, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States